CLINICAL TRIAL: NCT03719014
Title: A Prospective, Multi-Center, Non-randomized, Single Arm, Open Label, Pivotal Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions
Brief Title: Cohort B of the Pivotal Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nitiloop Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CLP-01 Cohort B
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Coronary Occlusion
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Intervention Model Description: This is an open label, multi-center, prospective, supplemental study in which the device, NovaCross™ CTO micro-catheter, will be tested in up to 60 patients scheduled to undergo CTO-PCI using an anterograde approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NovaCross (Experimental): the NovaCross is a guidewire positioning and support micro-catheter for improving chronic total occlusion (CTO) crossability. The NovaCross gains its supportive characteristics through the use of a unique operator-controlled Nitinol scaffold and an extandable segment, both at its distal tip.
  Interventions: Device: NovaCross

INTERVENTIONS:
Device: NovaCross — The NovaCross micro-catheter will be used during a standard of care Percutanous Coronary Intervention (PCI) on subjects diagnosed with at least one coronary chronic total occlusion (CTO), in order to assist the operator in guidewire stability and centralization.

SUMMARY:
A Prospective, Multi-Center, Non-randomized, Single arm, Open label, Supplemental Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 25-80
* Patient understands and has signed the study informed consent form
* Patient has an angiographic documented Chronic Total Occlusion (i.e. >3 months occlusion duration) showing distal TIMI flow 0, with a reference diameter of at least 2 millimeters.
* Left ventricle ejection fraction > 25%

Exclusion Criteria:

* Patient unable to give informed consent.
* Elevated CK-MB or troponin at baseline
* Patient is known or suspected not to tolerate the contrast agent
* Chronic Total Occlusion is located in aorto-ostial location, SVG CTO, in-stent occlusion
* Appearance of a fresh thrombus or intraluminal filling defects
* Intolerance to Aspirin and/or inability to tolerate a second antiplatelet agent (Clopidogrel and Prasugrel and Ticagrelor)
* Cardiac intervention within 4 weeks of the procedure
* Severe renal insufficiency with eGFR<30 ml/min/1.72 m2
* Congestive heart failure [New York Heart Association (NYHA) Class III\IV] CSA Class IV
* Life expectancy < 2 years due to other illnesses
* Acute or unstable medical disorder/disease that may cause a risk to patient, including:

  i. Recent myocardial infarction (MI) (within the past two weeks) ii. Significant anemia (e.g. hemoglobin < 8.0 mg / dl) iii. Recent major cerebrovascular event (history of stroke or TIA within 1 month) iv. Severe uncontrolled systemic hypertension (e.g., >180/100 mmHg) v. Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Measure - Rate of in-hospital MACE events | up to 30 days
  Defined as the composite of death, myocardial infarction (MI), or urgent revascularization (target vessel revascularization (TVR) or urgent coronary artery bypass surgery (CABG)).
Primary Outcome Measure - Intra-procedural technical succees | Intra-procedure
  Intra-procedural technical success defined as the ability of the NovaCross™ microcatheter to successfully facilitate placement of a guidewire beyond a native coronary chronic total occlusion (CTO) in the true vessel lumen

SECONDARY OUTCOMES:
Outcome Measure - Rate of procedure success | Procedure
  The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion, and place a coronary stent with residual lumen stenosis of less than 30% while restoring antegrade TIMI 3 flow
Outcome Measure - Technical adaptation of the Micro-catheter to the guidewire | Procedure
  The ability of the NovaCross™ micro-catheter to facilitate a guidewire successfully penetrating the proximal cap of the CTO
Outcome Measure - Effective micro-catheter crossability | Procedure
  The effectiveness of the extendable portion in intra-CTO microcatheter crossability
Outcome Measure - Ease of Use | Procedure
  Operator's ability to visualize the NoveCross micro-catheter throughout the procedure, as well as to assess the ease of use of the NovaCross
Safety Measure - Myocardial Infraction (MI) rate | up to 30 days
  Rate of MI events, as defined according to the SCAI and 3rd universal definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walsh, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (3):
- United States (3):
  - Little Rock Medical Center, Little Rock, Arkansas
  - Nyph/Cumc, New York, New York
  - York Hospital, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No